CLINICAL TRIAL: NCT02878486
Title: Intervention to Reduce Sitting Time in Mild Cognitive Impairment
Brief Title: Intervention to Reduce Sedentary Time
Acronym: ReST-MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Amber Watts, PhD, Assistant Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003981
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Physical activity; Alzheimer's disease; cognitive impairment; sedentary behavior; insulin sensitivity
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Alzheimer Disease; Sedentary Behavior; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Subjects will have clinic visits, home visits, and telephone visits. Subjects will be asked to wear a wrist monitor (Jawbone Up) for duration of the study, will meet with the study team to review Physical Activity Education and also be asked to wear the ActivPAL device to assess sitting time.
  Interventions: Device: Jawbone Up; Behavioral: Physical Activity Education; Device: ActivPAL
- Group 2 (Active Comparator): Subjects will make clinic visits. At home visits, subjects will meet with the study team to review Physical Activity Education and also be asked to wear the ActivPAL device to assess sitting time.
  Interventions: Behavioral: Physical Activity Education; Device: ActivPAL

INTERVENTIONS:
Device: Jawbone Up — Jawbone Up is a wrist wore water resistant activity monitor.
  Arms: Group 1
Behavioral: Physical Activity Education — A study team member will discuss benefits of changing sitting habits and ways to make changes to personal habits.
Device: ActivPAL — Devices measures postural changes over time. Participants will wear device for 7 days. The device measures time sitting, standing, and posture changes (i.e. sit-to-stand).

SUMMARY:
The purpose of this study is to determine whether the researchers can help people change the amount of time they spend in sitting activities and whether this change might improve health outcomes.

DETAILED DESCRIPTION:
Specific Aim 1: Determine feasibility of a 12-week home and telephone based intervention in older adults with mild cognitive impairment targeting both the impaired individual and their study partner to help initiate and maintain behavior change. We will recruit KUADC registry participants with MCI and their caregivers (as study partners). Behavioral interventions are more effective when there is built in social support. We will evaluate feasibility in terms of successful recruitment and retention of participants, 10% or less of technological failures, rate of participant concerns addressed by phone and at home visits, acceptability of the intervention to participants (measured by questionnaires during home visits).

Specific Aim 2: Determine whether a 12-week home and telephone based intervention results in reduced total sitting time and shorter bouts of sitting in older adults with MCI and their caregivers. Electronic postural monitors will record sitting time for a duration of one week at three time points (pre-intervention, mid-intervention, and post-intervention). The intervention includes 1) feedback from baseline monitoring, 2) educational and goal setting session with the participants and research staff, 3) wrist worn monitors that alert wearers to sitting times >30 minutes, 4) home and telephone visits to address physical, psychological, and home environment barriers to behavior change. Changes in sitting time and breaks from sitting will be compared between baseline, mid-intervention, and post-intervention measurement occasions.

Specific Aim 3: Determine whether sedentary behavior intervention results in improved insulin sensitivity and glycemic control. To evaluate whether reduced sitting results in meaningful metabolic changes, we will measure postprandial insulin and glucose, and body composition, and evaluate changes from pre- to post- intervention adjusting for relevant covariates.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the University of Kansas (KU) Alzheimer's Disease Center (ADC) Registry
* Clinical Dementia Rating (CDR) = 0.5
* Inactive status as determined by the Measure of Older Adults' Sedentary Time (MOST) questionnaire
* Retired or <20 hours/week in an office
* Lives with partner in a community dwelling setting

Exclusion Criteria:

* Unable to stand or walk unassisted
* Inadequate visual, auditory, or English language capacity
* Adhesive allergy
* Current uncontrolled Type 2 diabetes
* Unwilling to change sitting behavior

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Watts, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group (Jawbone Up Wrist Monitor): Subjects will have clinic visits, home visits, and telephone visits. Subjects will be asked to wear a wrist monitor (Jawbone Up) for duration of the study, will meet with the study team to review Physical Activity Education and also be asked to wear the ActivPAL device to assess sitting time.
  Jawbone Up: Jawbone Up is a wrist wore water resistant activity monitor.
  Physical Activity Education: A study team member will discuss benefits of changing sitting habits and ways to make changes to personal habits.
  ActivPAL: Devices measures postural changes over time. Participants will wear device for 7 days. The device measures time sitting, standing, and posture changes (i.e. sit-to-stand).
- Control Group (No Wrist Monitor): Subjects will make clinic visits. At home visits, subjects will meet with the study team to review Physical Activity Education and also be asked to wear the ActivPAL device to assess sitting time.
  Physical Activity Education: A study team member will discuss benefits of changing sitting habits and ways to make changes to personal habits.
  ActivPAL: Devices measures postural changes over time. Participants will wear device for 7 days. The device measures time sitting, standing, and posture changes (i.e. sit-to-stand).
Period: Overall Study
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group (Jawbone Up Wrist Monitor): Intervention group will have vibrotactile reminders from a wrist worn device, education about changing sitting habits, and coaching to change habits
- Control Group (No Wrist Monitor): Control group will have education about changing sitting habits, no coaching or vibrotactile reminders
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.33 (8.62) | 80.83 (5.35) | 81.08 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Sitting Time
Description: Average daily sitting time (minus sleep) at 6 weeks minus average daily sitting time (minus sleep) at baseline measured using the activPAL monitor
Time Frame: Change from Baseline to Week 6
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Number analyzed (Participants) | 3 | 3
minutes per day | 0.43 (0.53) | 0.98 (1.82)

2. Secondary Outcome: Change in Average Daily Sitting Time
Description: Average daily sitting time (minus sleep) at 12 weeks minus average daily sitting time (minus sleep) at baseline measured using the ActivPAL monitor
Time Frame: Change from Baseline to Week 12
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Number analyzed (Participants) | 3 | 3
minutes per day | -0.17 (0.41) | -0.24 (0.56)

3. Secondary Outcome: Number of Sitting Bouts Greater Than 30 Min
Description: Change in the number of sitting bouts greater than 30 min measured using the ActivPAL monitor
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: sitting bouts
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Number analyzed (Participants) | 3 | 3
sitting bouts | 1 (1.41) | .167 (.764)

4. Secondary Outcome: Change in Glucose Levels Area Under the Curve in Response to Mixed Meal Tolerance Test
Description: The average area under the curve at week 12 minus the average area under the curve at baseline. Blood was collected at baseline (pre-mixed meal). Post-mixed meal it was collected at 15, 30, 45, 60, 90, 120 minutes. The Area Under the Curve (AUC) was computed using the trapezoidal rule as we have previously described (Burns et. al. 2012, Morris et al 2014). This results in a single AUC pre-intervention value, and a single AUC post-intervention value for each metabolic outcome measure (glucose, insulin, etc).
  The Area Under the Curve (AUC) for each individual is calculated as a single unitless value that results from calculating the definite integral under a timecourse curve. This method has been widely used and cited in metabolic studies for more than two decades https://doi.org/10.2337/diacare.17.2.152. This results in a single unitless AUC pre-intervention value, and a single AUC post-intervention value for each metabolic outcome response measure (glucose, insulin, etc).
Time Frame: Change from Baseline to Week 12
Population: Only three participants had data available for the mixed meal tolerance test
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Number analyzed (Participants) | 2 | 1
unitless | 178.88 (2144.12) | 1008.38 (0)

5. Secondary Outcome: Change in Insulin Levels Area Under the Curve Based on a Mixed Meal Tolerance Test
Description: as for outcome 4
Time Frame: Change from Baseline to Week 12
Population: Only three participants had data available for the mixed meal tolerance test
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Number analyzed (Participants) | 2 | 1
unitless | 2623.43 (1929.77) | 1776.38 (0)

6. Post Hoc Outcome: Change in HOMA-IR (Homeostatic Model Assessment of Insulin Resistance)
Description: HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) is calculated as fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. The average HOMA-IR at week 12 minus the average HOMA-IR at baseline. A lower score means a person is more sensitive to insulin, whereas a higher score indicates greater resistance to insulin. The HOMA-IR is a tool for calculating degree of insulin resistance. Given that this is a product of insulin and glucose values divided by a constant, there is no maximum score for this measure. The minimum score would be zero as neither insulin or glucose would drop below zero.
Time Frame: Change from baseline to week 12
Population: Only three participants had data available for the mixed meal tolerance test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group (Jawbone Up Wrist Monitor) | Control Group (No Wrist Monitor)
Number analyzed (Participants) | 2 | 1
units on a scale | 96438.33 (25698.46) | 63383.80 (0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Note that only 3 of the 6 participants were tested with the mixed meal tolerance test and blood draws. Thus, only 3 were exposed to potential risks associated with these procedures.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1 (N=3) | Group 2 (N=3)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rash at the site of adhesive used to attach monitoring device
IV site irritation (Skin and subcutaneous tissue disorders) | 1/2 (1) | 0/1 (0) — skin irritation at the site of IV used for blood collection

LIMITATIONS AND CAVEATS:
This is a very small sample and results are not generalizeable. It is a pilot study for feasibility only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT02878486/Prot_SAP_000.pdf